CLINICAL TRIAL: NCT04313816
Title: Difference Between Patient Vaccine Hesitancy and Perception by Their Family Physician of Their Vaccine Hesitancy
Acronym: DiffHésiVac
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.288; 2019-A02487-50 (Other: ID RCB)
Record Dates: First submitted 2020-01-14; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Vaccine Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- unique group: patients visiting their family physician
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — no intervention at all apart from filling a brief questionnaire
  Other Names: no intervention at all apart from filling a brief questionnaire

SUMMARY:
The investigators will ask to a patient and his/her family physician to complete in parallel a brief questionnaire at the beginning of the consultation:

* for the patient: self-evaluation of his/her vaccine hesitancy (with a 0-100 scale)
* for the physician: evaluation of this patient vaccine hesitancy (on the same 0-100 scale) Each of these 2 questionnaires should be filled blindly from the other.

DETAILED DESCRIPTION:
The investigators will ask to a patient and his/her family physician to complete in parallel a brief questionnaire at the beginning of the consultation:

* for the patient: self-evaluation of his/her vaccine hesitancy (with a 0-100 scale)
* for the physician: evaluation of this patient vaccine hesitancy (on the same 0-100 scale) Each of these 2 questionnaires should be filled blindly from the other.

The investigators will recruit 400 to 500 patients in 20 medical practices of general practioners.

ELIGIBILITY:
Inclusion Criteria:

* visiting the family physician
* accepting the study after information

Exclusion Criteria:

* none apart from the reverse of inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients visiting their family physician in one participating medical practice
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
difference between patient's vaccine hesitancy and perception by his/her family physician of his/her vaccine hesitancy. | one day
  Each participant will evaluate hi/her vaccine hesitancy on a 0-100 scale; his/her family physician will also evaluate the vaccine hesitancy of this participant on the same 0-100 scale.
  The outcome 1 is the difference between patient's vaccine hesitancy and perception by his/her family physician of his/her vaccine hesitancy (on this 0-100 scale).
  These are arbitrary units.

CONTACTS AND LOCATIONS:
Locations (1):
- EPAULARD, Grenoble, France

IPD SHARING:
Plan to Share IPD: No
non sharing of individual data.